CLINICAL TRIAL: NCT04993495
Title: Prospective Observational Study Evaluating the Potential Impact of a Hemorrhagic Risk Stratification Score in Patients With Mild Head Trauma
Brief Title: Study Evaluating the Potential Impact of a Hemorrhagic Risk Stratification Score in Patients With Mild Head Trauma
Acronym: TCL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC21_0140
Record Dates: First submitted 2021-07-22; First posted 2021-08-06 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-07

CONDITIONS: Head Injury Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head injuries are a common reason for consultation in emergency departments. The clinical severity of head injury is assessed using the Glasgow Coma Scale (GCS). Between 71% and 97.5% of patients with head trauma seen in the emergency department are considered minor, that is to say with an initial GCS 13 and the consequences are quite variable. Three to 10% of patients will have short, medium or long-term health consequences. According to the studies, there are between 2.1 and 8% of intracranial bleeding immediate or delayed (up to one month), with about 1% of them, the need to resort to neurosurgery.

Following a minor head trauma, it is recommended, in the absence of clinical signs of severity, to realize a brain scan (cerebral computerized tomography scan (CT scan): reference imaging examination) within 6h (between 4 hours and 8 hours according to studies), a hospital surveillance of 24h, with the realization of a control scanner within 12 hours to 24 hours in case of treatment by anticoagulants or antiaggregation.

In December 2015, Journal of the American Medical Association published an article evaluating two clinical algorithms across the Atlantic, the New Orleans Criteria (NOC) and the Canadian CT Head Rule, to identify a group of patients with a very low risk of severe brain damage.

The performance of this score is unquestionably, however, it does not include patients treated with antiplatelet or anticoagulant drugs; risk factors having a decisive impact on the incidence of intracranial bleeding.

In this context, various studies have been carried out retrospectively in Angers to assess the incidence and risk factors of the occurrence of an immediate or delayed intracerebral hemorrhage in patients with minor head trauma with or without anti-thrombotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18 years old
* head injury
* Glasgow Coma Scale > or = 13

Exclusion Criteria:

* Refusal of participation,
* Indication of a scanner for a reason other than minor head injury
* follow-up not possible
* pregnant woman or breastfeeding
* patients in life-threatening emergency situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the emergency department for minor head injury
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-07-07 (Estimated); Study Completion 2023-07-07 (Estimated)

PRIMARY OUTCOMES:
intracranial hemorrhage rate in patients in patients considered to be low risk according to the score created by hospital of Angers (negative predictive value). | Day 30
  to assess stratification score performance to predict the occurrence of acute intracranial bleeding in patients with minor head injury

SECONDARY OUTCOMES:
loss of one point on the rankin scale | Day 30
  Performance assessment of hemorrhagic risk stratification score to predict severe intracerebral hemorrhage
number of cerebral computerized tomography scan | Day 30
  Assessment of the potential reduction in the number of scanners if the score had been applied.
time spent in emergencies | Day 1
  Retrospective assessment of the potential impact of applying the score on the length of time spent in emergencies

CONTACTS AND LOCATIONS:
Locations (1):
- DOUILLET Delphine, Angers, France